CLINICAL TRIAL: NCT02310269
Title: Non-interventional Study for the Generation of Long Term Safety and Efficacy Data of Pasireotide s.c. in Patients With Cushing's Disease (Post-Authorization Safety Study)
Brief Title: Long Term Safety and Efficacy of Pasireotide s.c. in Patients With Cushing's Disease
Status: Completed | Type: Observational
Sponsor: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Other Study IDs: CSOM230B2410
Record Dates: First submitted 2014-09-26; First posted 2014-12-08 (Estimated); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-07

CONDITIONS: Cushings Disease
Keywords: Cushing's disease,; pasireotide s.c.; Signifor
MeSH Terms: conditions — Adrenocortical Hyperfunction; Pituitary ACTH Hypersecretion | interventions — pasireotide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1/new use cohort: Subjects who initiated pasireotide s.c. at time of study entry (on or after the signing of the informed consent or acknowledging an equivalent document -for example, written information- as per country regulation).
  Interventions: Drug: Pasireotide
- Cohort 2/prior use cohort: Subjects who initiated pasireotide s.c. prior to study entry.
  Interventions: Drug: Pasireotide

INTERVENTIONS:
Drug: Pasireotide
  Other Names: Signifor

SUMMARY:
This is a non-interventional, multinational, multi-center post-marketing study, to further document the safety and efficacy of pasireotide s.c. administered in routine clinical practice in patients with Cushing's disease. Patients with Cushing's disease and treated with pasireotide s.c. alone and in combination with other therapies will be monitored. For this study, each enrolled patient will be followed up for 3 years after enrollment. Patients who permanently discontinue pasireotide s.c. prior to completing the 3-year observation period will be followed up for 3 months after the last dose of pasireotide s.c.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent or equivalent document (e.g., written information) as per country regulation prior to registration of any patient data
* Male or female patients aged 18 years or older with a diagnosis of Cushing's disease for whom surgery has failed or for whom surgery is not an option
* Patients must be treated with pasireotide s.c. started either at the first visit for this study or prior to study entry

Exclusion Criteria:

* Patients with ectopic ACTH-dependent Cushing's syndrome
* Patients with adrenal Cushing's syndrome
* Patients with Pseudo Cushing's syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population will consist of male and female patients aged 18 years or older with a diagnosis of Cushing's disease for whom surgery has failed or for whom surgery is not an option and who are treated with pasireotide s.c.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2013-03-28 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario MALDONADO, MD, Study Director — Recordati AG
Locations (54):
- United States (7):
  - St Josephs Hospital and Medical Center, Phoenix, Arizona
  - University of Southern California CSOM230B2410 - SC, Los Angeles, California
  - Massachusetts General Hospital SC - SOM230B2410, Boston, Massachusetts
  - Ohio State University SC - SOM230B2410, Columbus, Ohio
  - Endocrinology Services, Bend, Oregon
  - Allegheny Endocrinology Associates, Pittsburgh, Pennsylvania
  - Swedish Medical Center Dept.ofSeattle Neuroscience(2), Seattle, Washington
- Canada (3):
  - Centre de recherche du CHUM CRCHUM, Montreal, Quebec
  - CHUL Centre de recherche du CHU, Québec, Quebec
  - CHUS - Hopital Fleurimont, Sherbrooke, Quebec
- Centro Medico Imbanaco de Cali, Cali, Colombia
- France (9):
  - CHU Amiens Picardie Site Nord, Amiens
  - HCL-Groupe Hospitalier Est, Bron
  - Recordati Investigative Site, Lille
  - AP-HM - Hopital de la Conception, Marseille
  - Hopital Lapeyronie, Montpellier
  - Hopital Cochin, Paris
  - Hopital Robert Debre, Reims
  - HIA Begin, Saint-Mandé
  - CHU de Saint Etienne, Saint-Priest-en-Jarez
- Germany (14):
  - Universitaetsklinikum Aachen, Aachen
  - Universitaetsmedizin Charite, Berlin
  - Univ.-Klinikum Düsseldorf, Düsseldorf
  - Universitaetsklinikum Erlangen Nuernberg, Erlangen
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Praxis Dr.med.Frank Ackermann, Halle
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Universitaetsklinikum Leipzig AoR, Leipzig
  - Universitaetsklinikum Magdeburg AoR, Magdeburg
  - Universitaetsklinikum Muenchen LMU, München
  - Medicover Muenchen Ost MVZ, München
  - Praxis Michael Droste, Oldenburg
  - Universitaetsklinikum Wuerzburg, Würzburg
- Israel (2):
  - Rabin Medical Centre Belinson, Petah Tikva
  - Tel Aviv Sourasky Medical Centre Ichilov, Tel Aviv
- Italy (9):
  - AOU Osp Riuniti Umberto I GM Lancisi G Salesi Univ Studi, Ancona, AN
  - Az.Ospe.Universitaria Policlinico G. Martino Univ.di Messina, Messina, ME
  - Fond IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan, MI
  - Stab.Osp.S.Luca P.O. S.Luca-S.Michele-Ist.Auxol. Italiano, Milan, MI
  - Az Osp Univ Policlinico P Giaccone Universita Studi Palermo, Palermo, PA
  - Azienda Ospedaliera di Padova Universita degli Studi, Padua, PD
  - Az Ospedaliero Universitaria Pisana Pres Osped di Cisanello, Pisa, PI
  - P O Molinette AO Citta della Salute e della Scienza Torino, Torino, TO
  - O Universitaria Policlinico Federico II Univ Studi Fed II, Napoli
- Hotel Dieu de France Hospital, El Achrafiyé, Lebanon
- Netherlands (2):
  - Maastricht Universitair Medisch Centrum, Maastricht, AZ
  - Radboudumc, Nijmegen
- Romania (4):
  - Spitalul Clinic Judetean de Urgenta Brasov, Brasov
  - Institutul de Endocrinologie "I. C. Parhon", Bucuresti, Bucharest
  - Spitalul Clinic Jude Emergency Clinical County Hospital Cluj, Cluj-Napoca
  - County Hospital Tg. Mures, Târgu Mureş
- United Kingdom (2):
  - Derriford Hospital, Plymouth
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Manetti L, Deutschbein T, Schopohl J, Yuen KCJ, Roughton M, Kriemler-Krahn U, Tauchmanova L, Maamari R, Giordano C. Long-term safety and efficacy of subcutaneous pasireotide in patients with Cushing's disease: interim results from a long-term real-world evidence study. Pituitary. 2019 Oct;22(5):542-551. doi: 10.1007/s11102-019-00984-6. PMID 31440946

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects: Patients with Cushing's disease and treated with pasireotide s.c. alone and in combination with other therapies.
Period: Overall Study
Arm/Group | All Subjects
Started | 152
Completed | 29
Not Completed | 123

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (13.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 126
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 118
  More than one race | 0
  Unknown or Not Reported | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability Profile of Pasireotide s.c.
Description: Number of pasireotide s.c related adverse events and serious adverse events, when administered as monotherapy or in combination with other therapies in patients with Cushing's disease
Time Frame: 3-year follow-up
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1/New Use Cohort: Subjects who initiated pasireotide s.c. at time of study entry (on or after the signing of the informed consent or acknowledging an equivalent document -for example, written information- as per country regulation).
  Pasireotide
- Cohort 2/Prior Use Cohort: Subjects who initiated pasireotide s.c. prior to study entry.
  Pasireotide
Arm/Group | Cohort 1/New Use Cohort | Cohort 2/Prior Use Cohort
Number analyzed (Participants) | 43 | 105
Participants
  At least 1 treatment-emergent SAE that was suspected to be pasireotide-related. | 11 | 13
  A treatment-emergent AE of any grade that was suspected to be pasireotide-related. | 34 | 54

ADVERSE EVENTS:
Time Frame: Adverse events and Serious Adverse Events will be followed-up and collected from patient's enrollment into the study until 28 days after the last dose of pasireotide s.c. at the patient's last follow-up visit. Adverse events and Serious Adverse Events will be collected until 3 months after the last dose for patients who permanently discontinue pasireotide s.c. prior to completing 3-year observation period.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 5/148
Serious Adverse Events (participants affected / at risk) | 49/148
Other Adverse Events (participants affected / at risk) | 132/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=148)
Hyperglycaemia (Metabolism and nutrition disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 3
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 6
Metabolic alkalosis (Metabolism and nutrition disorders) | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 2
Cerebral haematoma (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
IIIrd nerve paresis (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 3
Pituitary-dependent Cushing's syndrome (Endocrine disorders) | 3
Hyperadrenocorticism (Endocrine disorders) | 2
Adrenocortical insufficiency acute (Endocrine disorders) | 1
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1
Drug ineffective (General disorders) | 4
General physical health deterioration (General disorders) | 3
Asthenia (General disorders) | 1
Fatigue (General disorders) | 1
Malaise (General disorders) | 1
Pneumonia (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 2
COVID-19 (Infections and infestations) | 1
Meningitis haemophilus (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pyonephrosis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Atrial fibrillation (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Cortisol increased (Investigations) | 7
Hepatic enzyme increased (Investigations) | 2
CSF test abnormal (Investigations) | 1
Cortisol free urine increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Grip strength decreased (Investigations) | 1
Transaminases increased (Investigations) | 1
Weight decreased (Investigations) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Gastrointestinal hypermotility (Gastrointestinal disorders) | 1
Tooth disorder (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 4
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pituitary cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Stress fracture (Injury, poisoning and procedural complications) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Calculus urinary (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Confusional state (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Visual impairment (Eye disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2.7% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=148)
Nausea (Gastrointestinal disorders) | 38
Diarrhoea (Gastrointestinal disorders) | 23
Diabetes mellitus (Metabolism and nutrition disorders) | 19
Hyperclycaemia (Metabolism and nutrition disorders) | 18
Asthenia (General disorders) | 16
Fatigue (General disorders) | 16
Headache (Nervous system disorders) | 16
Adrenal Insuffiency (Endocrine disorders) | 12
Abdominal pain (Gastrointestinal disorders) | 11
Cholelithiasis (Hepatobiliary disorders) | 11
Hypertension (Vascular disorders) | 11
Drug Ineffective (General disorders) | 10
Vomiting (Gastrointestinal disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Dizziness (Nervous system disorders) | 8
Nasopharyngitis (Infections and infestations) | 8
Hyperadrenocorticism (Endocrine disorders) | 7
Hypercholesterolemia (Metabolism and nutrition disorders) | 7
Hypoglycaemia (Metabolism and nutrition disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Vertigo (Nervous system disorders) | 6
Hepatic Steatosis (Hepatobiliary disorders) | 5
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 5
Feeling cold (General disorders) | 4
Hypothyroidism (Metabolism and nutrition disorders) | 4
Weight decreased (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Physician or Institution must submit to Sponsor at least 45 days before any publication, the material that they would publish, for Sponsor review and approval of this publication.

DOCUMENTS (2):
  • Study Protocol (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/69/NCT02310269/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT02310269/SAP_001.pdf